CLINICAL TRIAL: NCT02278640
Title: Prospective, Multicenter, Study Evaluating Vessel Sealing Utilizing the Harmonic ACE®+7 Shears During Total Laparoscopic Hysterectomy
Brief Title: Harmonic ACE®+7 Shears in Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENG-14-002
Record Dates: First submitted 2014-10-10; First posted 2014-10-30 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-07

CONDITIONS: Benign Disease Where Total Hysterectomy is Indicated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Harmonic ACE®+7 Shears (Other): Single Arm study using Harmonic ACE for dissection and transection in Hysterectomy
  Interventions: Device: Harmonic ACE®+7 Shears

INTERVENTIONS:
Device: Harmonic ACE®+7 Shears — Vessel/pedicle sealing performance assessed for transection and sealing of the of the uterine vasculature.

SUMMARY:
This is a prospective, non-randomized, single arm, multicenter, study to assess the initial clinical experience with the Harmonic ACE®+7 Shears by evaluating vessel sealing during total laparoscopic hysterectomy. The study will not modify or influence current surgeon technique. Investigators will perform each procedure using the device in compliance with their standard surgical approach and product labeling.

The Harmonic ACE®+7 Shears is cleared for commercial distribution and will be used in accordance with approved product labeling. The Harmonic ACE®+7 Shears will be assembled, calibrated, and/or used in accordance with manufacturer design specifications, product instructions and guidelines

DETAILED DESCRIPTION:
Study Population: Subjects enrolled into this study will undergo elective total laparoscopic hysterectomy for benign indications wherein dissection and transection of the uterine vasculature is indicated.

Primary Variables: Percentage of subjects achieving hemostasis at the named vessel/pedicle (UA or UP) on the left side. Percentage of subjects achieving hemostasis at the named vessel/pedicle (UA or UP) on the right side.

Definition: Hemostasis of the named vessel or pedicle is a dichotomous variable (i.e. yes or no). "Yes" is defined as the hemostatic transection of the uterine vasculature (left / right) with at least one use of the device in Advanced Hemostasis mode (a completed cycle with the second activation tone heard) without the use of additional hemostatic measures (i.e. tissue sealers, cautery devices, hemoclips, staples, sutures, fibrin sealants, etc.) other than the Harmonic ACE®+7 device.

Note: Multiple applications of the Advanced Hemostasis mode and/or additional applications of the device in a maximum (MAX) or minimum (MIN) mode are allowed.

Secondary Endpoints:

Percentage of subjects achieving hemostasis at the OP on the left and/or right side.

If the study procedure also includes the transection and sealing of one or both OPs, hemostasis of the left and/or right OP will also be recorded. Hemostasis of the OP is a dichotomous variable (i.e. yes or no). "Yes" is defined as the hemostatic transection of the ovarian vasculature (left and/or right) with at least one use of the device in Advanced Hemostasis mode (a completed cycle with the second activation tone heard) without the use of additional hemostatic measures (i.e. tissue sealers, cautery devices, hemoclips, staples, sutures, fibrin sealants, etc.).

Note: Multiple applications of the Advanced Hemostasis mode or the device in a MAX or MIN mode are allowed.

Exploratory endpoints include:

Requirement for additional measures to obtain hemostasis on the named vessel/pedicle (UA or UP and/or OP) on the left and right side Use of other energy devices (tissue sealers, cautery devices) - Graded as yes or no; if "yes", the name and type, time of application (24 hour clock).

Use of additional hemostatic products (e.g. hemoclips, staples, sutures, fibrin sealants) - Graded as yes or no; if "yes", the name and type, number/volume, and time of application (24 hour clock).

Complications associated with vaginal cuff healing including dehiscence or separation, infection, cellulitis, abscess, inflammation, and granulation associated with each suture used as part of the study.

Adverse events attributed to the study device or procedure will be collected from time of surgery to Visit 4 (Approximately 4 to 6 weeks after study surgery or as per standard of care (SOC)).

No formal sample size determination is required for this study. Approximately 40 subjects from the United States and the European Union are planned to be enrolled into this study.

Global indication for use of the The Harmonic ACE®+7, 5mm Diameter Shears with Advanced Hemostasis:

Indicated for soft tissue incisions when bleeding control and minimal thermal injury are desired. The instruments can be used as an adjunct to or substitute for electrosurgery, lasers and steel scalpels in general, plastic, pediatric, gynecologic, urologic, thoracic, exposure to orthopedic structures (such as spine and joint space), sealing and transection of lymphatic vessels, and other open and endoscopic procedures. The instruments allow for the coagulation of vessels up to and including 7mm in diameter, using the Advanced Hemostasis function.

ELIGIBILITY:
Inclusion Criteria:

Subjects satisfying all of the following criteria will be considered the screening population and will be eligible for participation in this study:

1. Indicated for elective total laparoscopic hysterectomy
2. Age >=40 years and no future desire for fertility

Exclusion Criteria:

Subjects with any of the following criteria will be excluded from the study:

Preoperative exclusion criteria:

1. Known or suspected uncontrolled bleeding disorders
2. Subjects unlikely to comply with protocol procedures or adhere to the study visit schedule
3. Any condition rendering a subject unable to understand the nature, scope, and possible consequences of the study or study procedures
4. Any Subject unwilling to sign the study informed consent document
5. Any suspected malignancy
6. Any Subject of childbearing potential with a positive or serum pregnancy test within 24 hours prior to surgery

   Intra-operative exclusion criteria:
7. Any intra-operative findings identified by the surgeon that may preclude conduct of the study procedure

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Florida Hospital Celebration Health, Celebration, Florida
  - The Advanced Gynecological Surgery Institute, Schaumburg, Illinois
- Gynaecoloog (aandachtsgebied: endoscopische chirurgie), Nijmegen, Netherlands
- The Royal Surrey County Hospital NHS Trust, Surrey, United Kingdom

REFERENCES:
- [Background] Nieboer TE, Steller CJ, Hinoul P, Maxson AJ, Schwiers ML, Miller CE, Coppus SF, Kent AS. Clinical utility of a novel ultrasonic vessel sealing device in transecting and sealing large vessels during laparoscopic hysterectomy using advanced hemostasis mode. Eur J Obstet Gynecol Reprod Biol. 2016 Jun;201:135-9. doi: 10.1016/j.ejogrb.2016.03.035. Epub 2016 Apr 14. PMID 27124666

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Harmonic ACE®+7 Shears
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Set - all subjects in whom the procedure was started.
Arm/Group | Harmonic ACE®+7 Shears
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 39
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 15
  United States | 5
  United Kingdom | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Hemostasis at the Named Vessel/Pedicle (UA or UP) on the Left Side.
Description: Hemostasis of the named vessel or pedicle is a dichotomous variable (i.e. yes or no). "Yes" is defined as the hemostatic transection of the uterine vasculature (left / right) with at least one use of the device in Advanced Hemostasis mode (a completed cycle with the second activation tone heard) without the use of additional hemostatic measures (i.e. tissue sealers, cautery devices, hemoclips, staples, sutures, fibrin sealants, etc.) other than the Harmonic ACE®+7 device. Multiple applications of the Advanced Hemostasis mode and/or additional applications of the device in a maximum (MAX) or minimum (MIN) mode are allowed.
Time Frame: Intraoperative
Population: Safety Set - all subjects in whom the procedure was started.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Harmonic ACE®+7 Shears
Number analyzed (Participants) | 40
percentage of participants | 97.5 [86.8 to 99.9]

2. Primary Outcome: Percentage of Subjects Achieving Hemostasis at the Named Vessel/Pedicle (UA or UP) on the Right Side.
Description: as for outcome 1
Time Frame: Intraoperative
Population: Safety Set - all subjects in whom the procedure was started.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Harmonic ACE®+7 Shears
Number analyzed (Participants) | 40
percentage of participants | 92.5 [79.6 to 98.4]

3. Secondary Outcome: Percentage of Subjects Achieving Hemostasis at the Ovarian Pedicle on the Left Side.
Description: as for outcome 1
Time Frame: Intraoperative
Population: Safety Set With OP transection - All subjects in whom the procedure was started and for whom the transection of the ovarian pedicle was attempted.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Harmonic ACE®+7 Shears
Number analyzed (Participants) | 23
percentage of participants | 100.0 [85.2 to 100.0]

4. Secondary Outcome: Percentage of Subjects Achieving Hemostasis at the Ovarian Pedicle on the Right Side.
Description: as for outcome 1
Time Frame: Intraoperative
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Harmonic ACE®+7 Shears
Number analyzed (Participants) | 23
percentage of participants | 100.0 [85.2 to 100.0]

ADVERSE EVENTS:
Time Frame: Surgery to 4 weeks post surgery
Arm/Group | Harmonic ACE®+7 Shears
Serious Adverse Events (participants affected / at risk) | 3/40
Other Adverse Events (participants affected / at risk) | 23/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harmonic ACE®+7 Shears (N=40)
Haematoma infection (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harmonic ACE®+7 Shears (N=40)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 3 (3)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 2 (2)
Postoperative wound infection (Infections and infestations) | 2 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed that the first publication of results should be made in conjunction with the presentation of a joint, multicenter publication of the results with all PIs contributing data, analyses, and comments. If this publication was not submitted within 12 months after conclusion of the Study at all sites, or after Sponsor confirmed there would be no multicenter Study publication, whichever is first, the PIs could have published the results from their individual sites.